CLINICAL TRIAL: NCT05237765
Title: The Effect of Controlled Massage Applied at Birth on Labor Pain and Duration and Maternal Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Guluzar Sade, PhD Assistant Professor, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TarsusU
Record Dates: First submitted 2022-01-14; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Massage
Keywords: Birth, labor duration, labor pain, massage, satisfaction
MeSH Terms: conditions — Labor Pain; Personal Satisfaction | interventions — Control Groups; Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- midwife-controlled massage (Experimental)
  Interventions: Other: controlled (automatic) massage
- self-controlled massage (Experimental)
  Interventions: Other: controlled (automatic) massage
- control group (No Intervention)

INTERVENTIONS:
Other: controlled (automatic) massage — Massage methods that are performed with mechanical methods are called automated massage. Automated massage is also individual-controlled massage. This is because in automated massage, to relax, solve or reduce their pain, the individual applies the massage under their own control or under the control of someone else through a controller in a way where the duration and intensity of the massage in the body part of application vary. Individual-controlled massage devices may be in the form of chairs, cushions, beds and mattresses. These massage devices have functions such as vibrating, applying vacuum, imitating manual massage motions and applying heat.
  Arms: midwife-controlled massage; self-controlled massage

SUMMARY:
This study was carried out to determine the effect of controlled massage applied at birth on labor pain and duration and maternal satisfaction. The study was conducted as a randomized, controlled research. The research was conducted with 154 randomized pregnant women admitted to Erzurum Nenehatun Obstetrics and Maternity hospital between February-November 2019. The study consisted of 3 different groups: Group A included the pregnant women who received routine hospital care (control group n=53), Group B included the pregnant women who received midwife-controlled massage (n=50), and the Group C consisted of the pregnant women who received self-controlled massage (n=51). It was determined that the controlled massage intervention that was applied in this study reduced labor pain, but it did not affect the duration of labor or the satisfaction levels of the women.

DETAILED DESCRIPTION:
This study was conducted to determine the effects of controlled massage applied during labor on pain during labor, labor duration and maternal satisfaction. This was a randomized-controlled experimental study.The study was carried out with the participation of 154 randomly selected pregnant women at an Obstetrics and Gynecology Hospital located in a province in the Eastern Anatolia Region of Turkey between February and November 2019.The study included three groups (A: control group, B: midwife-controlled massage group, C: self-controlled massage group). The data were collected using a "Personal Information Form", the "Visual Analogue Scale (VAS)", the "Verbal Category Scale (VCS)", a "Partograph", an "Individual-Controlled Massage Follow-Up Form" and the "Scale for Maternal Satisfaction in Vaginal Delivery (SMSVD)".It was determined that the controlled massage intervention that was applied in this study reduced labor pain, but it did not affect the duration of labor or the satisfaction levels of the women.

IMPACT STATEMENT What is already known on this subject? Labor pain and outcomes occurring during labor are known and expected situation. Some nonpharmacological methods are applied to ensure that birth is easy and maternal satisfaction is high.

What the results of this study add? There is no studies using thecontrolled massage. In our study, it was found that controlled massage is effective on labor birth.

What the implications are of these findings for clinical practice and/or further research? Our study suggested that midwives and pregnant women could practice controlled massage to reduce labor pain.

ELIGIBILITY:
Inclusion Criteria:

* Having at least a primary school degree
* Not having a communication problem
* Having a primiparous term pregnancy (38-42 weeks)
* Not having an obstetric risk
* Being in the latent phase of labor (dilation 0-3cm)
* Having no contraindications for massage

Exclusion Criteria:

* Being multiparous
* Having a high-risk pregnancy
* Being in the active or transitional phase of labor
* Having a contraindication to massage

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | Delivery (when pregnant women come to the delivery room)
  This was a form that was prepared to collect information on the sociodemographic and obstetric characteristics of the participants. The form was filled when the pregnant woman was admitted to the labor room.
Visual Analogue Scale (VAS) | Latent, active and transition phase in labor
  The participants marked the levels of pain they perceived at the end of the latent, active and transitional phases of labor on a 10-cm ruler whose two extreme points represented "no pain at all" and "unbearable pain". This is a sensitive and reliable scale in the measurement of pain severity.
Verbal Category Scale (VCS) | Latent, active and transition phase of labor
  This is a one-dimensional, easy-to-apply and descriptive scale. The participants were asked to select one of the phrases "mild, uncomfortable, severe, highly severe, unbearable" that represented their pain status best.
Partograph | active and transition phase of labor
  It is a graphical form that is used starting with the active phase of labor and allows the detailed monitoring of the labor process and early detection of abnormal events. It was used in this study to determine the duration of labor based on its phases and the effect of the massage intervention on this duration.
Individual-Controlled Massage Follow-Up Form (ICMFF) | active and transition phase of labor
  ICMFF was a form that was developed by the researcher on which the active and transitional phases of labor were marked, and the duration and intensity of the massage that was applied were recorded by specifying the exact times. It was filled out by the researcher at the end of each massage application.
Scale for Maternal Satisfaction in Vaginal Delivery (SMSVD) | within a period of 1-4 hours postpartum
  This scale determines the satisfaction levels of mothers regarding the care they have received at the hospital in normal vaginal labor. It is a 5-point Likert-type (1: absolutely disagree to 5: absolutely agree) scale consisting of 43 items and 10 dimensions. Thirteen items in the scale are inversely scored. The scores of these 13 items are reversed while calculating the total score of the scale. Higher total scores indicate higher levels of maternal satisfaction from the care received at the hospital in the normal vaginal labor process. The cutoff point calculated for SMSVD is 150.5, where scores higher than 150.5 indicate high satisfaction levels, and those lower than 150.5 indicate low satisfaction levels. The form was applied by the researcher in the fourth phase of labor, when the mother was taken to her bed. The authors who developed the scale determined its Cronbach's alpha internal consistency coefficient as 0.91.

CONTACTS AND LOCATIONS:
Overall Officials: Gülüzar Sade, Dr., Principal Investigator — Tarsus University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)